CLINICAL TRIAL: NCT04850352
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel-design Clinical Study to Evaluate the Blood Triglyceride Decreasing Effect and Safety of Korean Post-Fermented Tea(Heukcha) Extracts
Brief Title: Clinical Study to Evaluate the Blood Triglyceride Decreasing Effect and Safety of Korean Post-Fermented Tea Extracts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amorepacific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: AP-PV-2018-02
Record Dates: First submitted 2021-04-14; First posted 2021-04-20 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Triglycerides High
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heukcha Extracts (Experimental): Take Heukcha Extracts capsule once daily for 8 weeks.
  Interventions: Dietary Supplement: Heukcha Extracts
- Placebo (Placebo Comparator): Take placebo capsule once daily for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Heukcha Extracts — Experimental group: Heukcha Extracts
  Arms: Heukcha Extracts
Dietary Supplement: Placebo — Placebo group
  Arms: Placebo

SUMMARY:
This study was conducted to investigate the effects of daily supplementation of Korean Post-Fermented Tea(Heukcha) Extracts on improvement of Blood Triglyceride Level.

DETAILED DESCRIPTION:
This study was a 8 week, randomized, multicenter, double-blind, placebo-controlled, parallel-design human trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 19 years old
* Who has fasting blood triglyceride levels ≥ 150 mg/dL
* Who voluntarily agreed to participate in the study and signed an informed consent form

Exclusion Criteria:

* Those who are taking functional food designed for dyslipidemia reduction within 4 weeks before study participation
* Those who have been diagnosed and are on medication with dyslipidemia, cardiovascular disease, kidney disease, liver disease or thyroid disease within 4 weeks before study participation
* Fasting plasma glucose >126 mg/dL or treatment with medications including oral hypoglycemic agents or insulin
* Who has used or is expected to inevitably use prohibited concomitant medications during the study
* Women who is pregnant /breast-feeding, or who has childbearing potential and does not use available contraceptives
* Who has dosed other study medications within 30 days before screening
* Who is determined ineligible for study participation by investigators for any other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in fasting triglycerides | Baseline, Week 4 and Week 8

SECONDARY OUTCOMES:
Change in total cholesterol, LDL-C, HDL-C | Baseline, Week 4 and Week 8
Change in BMI (kg/m2) | Baseline, Week 4 and Week 8
Change in Waist circumference (cm) | Baseline, Week 4 and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Belong Cho, MD, PhD, Principal Investigator — Seoul National University
Locations (3):
- South Korea (3):
  - KangBuk Samsung Medical Center, Seoul
  - Seoul National University, Seoul
  - St. Vincent's Hospital, College of Medicine, The Catholic University of Korea, Suwon